CLINICAL TRIAL: NCT01834846
Title: Impact of Perivascular Tissue on Endothelial Function and Vessel Structure in Vein Grafts Used for Coronary Artery Bypass Grafting: A Prospective, Randomized Controlled Trial.
Brief Title: Impact of Perivascular Tissue on Endothelial Function in Coronary Artery Bypass Grafting
Acronym: IMPROVE-CABG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 090486
Record Dates: First submitted 2013-04-15; First posted 2013-04-18 (Estimated); Last update posted 2021-01-05 (Actual); Status verified 2020-12

CONDITIONS: Myocardial Ischemia
Keywords: comparative study; Cardiac Surgical Procedures
MeSH Terms: conditions — Myocardial Ischemia | interventions — Congresses as Topic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- no-touch (Experimental): no-touch technique of harvesting the saphenous vein graft for coronary artery bypass grafting
  Interventions: Procedure: no-touch
- conventional (Active Comparator): conventional technique of harvesting the saphenous vein graft for coronary artery bypass grafting
  Interventions: Procedure: conventional

INTERVENTIONS:
Procedure: no-touch — The saphenous vein is exposed by a longitudinal incision, and all visible side branches ligated. The vein is then isolated together with a pedicle of surrounding tissue and manually distended and stored in a combination of blood and saline using a syringe, according to standard procedure at St. Olav's Hospital.
  Arms: no-touch
Procedure: conventional — The saphenous vein is exposed by a longitudinal leg incision, skeletonized from surrounding tissue, and side branches ligated. The vein is removed from the leg immediately after dissection, manually distended and stored in a combination of blood and saline using a syringe, according to standard procedure at St. Olav's Hospital.
  Arms: conventional

SUMMARY:
The success of coronary artery bypass grafting is reliant on the quality of the grafts used. A new technique for harvesting veins used as grafts has been introduced. The study hypothesis is that veins harvested with this technique have an improved endothelial function.

ELIGIBILITY:
Inclusion Criteria:

* Isolated elective, primary CABG requiring cardiopulmonary bypass
* Left ventricular ejection fraction >35%
* at least one saphenous vein graft required as part of revascularization strategy

Exclusion Criteria:

* Acute or chronic inflammatory diseases
* Malignancies
* Pregnancy
* Previous cardiac surgery
* Serum creatinine >120 μmol/L
* Coagulopathy
* Insulin dependent diabetes mellitus
* Smoking during last 6 months
* Leg not suitable for No-touch vein harvesting as judged by the operator.
* Need for nitrates on operation day
* not receiving statins

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Graft function | 6 months
  Graft function as evaluated by coronary angiography in the first 60 out of 100 patients
Graft function | 5 years
  Graft function as evaluated by coronary angiography in all 100 patients

SECONDARY OUTCOMES:
Morphological appearance of vein graft | 6 months
  As measured by angiography follow-up in the first 60 out of 100 patients
Morphological appearance of vein graft | 5 years
  As measured by angiography follow-up in all 100 patients
Postoperative leg wound complications | 6 weeks
  The following measures will be assessed in the first 60 out of 100 patients:
  * Signs of infection
  * Wound dehiscence
  * Aesthetics
  * Cutaneous sensory loss
  * Wound discomfort
Postoperative complications related to cardiac surgery | Discharge, 6 weeks, 6 months
  Major adverse cardiac and cerebral events in the first 60 out of 100 patients
  * Postoperative complications
  * Reoperation
  * Sternal dehiscence
  * Mediastinitis
Postoperative complications related to cardiac surgery | 5 years
  Major adverse cardiac and cerebral events in all 100 patients
  * Postoperative complications
  * Reoperation
  * Sternal dehiscence
  * Mediastinitis

CONTACTS AND LOCATIONS:
Overall Officials: Dag Ole Nordhaug, md phd, Principal Investigator — Norwegian University of Science and Technology
Locations (1):
- Institute for Circulation and Imaging, Trondheim, Sør-Trøndelag, Norway

REFERENCES:
- [Result] Pettersen O, Wiseth R, Hegbom K, Nordhaug DO. Pedicled Vein Grafts in Coronary Surgery Exhibit Reduced Intimal Hyperplasia at 6 Months. J Am Coll Cardiol. 2016 Jul 26;68(4):427-9. doi: 10.1016/j.jacc.2016.04.058. No abstract available. PMID 27443441
- [Result] Pettersen O, Haram PM, Winnerkvist A, Karevold A, Wahba A, Stenvik M, Wiseth R, Hegbom K, Nordhaug DO. Pedicled Vein Grafts in Coronary Surgery: Perioperative Data From a Randomized Trial. Ann Thorac Surg. 2017 Oct;104(4):1313-1317. doi: 10.1016/j.athoracsur.2017.03.076. Epub 2017 Jun 23. PMID 28648540
- [Derived] Pettersen O, Pociask E, Malinowski KP, Slezak M, Hegbom K, Wiseth R, Nordhaug DO. Reproducibility of optical coherence tomography in vein grafts used for coronary revascularization. Cardiol J. 2020;27(5):518-523. doi: 10.5603/CJ.a2018.0139. Epub 2018 Nov 16. PMID 30444258